CLINICAL TRIAL: NCT02553096
Title: Adaptive Computerized COPD Exacerbation Self-management Support (ACCESS): A Randomized Controlled Trial
Brief Title: Exacerbation Self-management in COPD: The ACCESS Study
Acronym: ACCESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL49741 .091.14
Record Dates: First submitted 2015-08-05; First posted 2015-09-17 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: exacerbations; self-management support; software application
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: 2-block randomised trial
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACCESS (Experimental): ACCESS is used when participants experience more COPD symptoms.
  Interventions: Device: ACCESS
- paper plan (No Intervention): Paper exacerbation action plan is used when participants experience more COPD symptoms.

INTERVENTIONS:
Device: ACCESS — The ACCESS system consists of a smartphone, a pulse-oximeter, a spirometer and a forehead thermometer. Questions concerning changes in symptoms, physical limitations and emotions are answered by touch screen on the smartphone, complemented by measurements of the pulse-oximeter, spirometer and thermometer. Based on this information, the system calculates the current risk of an exacerbation and, when applicable, the participant will receive personalized instructions about which actions to take in order to manage the exacerbation. Participants are instructed to use ACCESS in case of symptom worsening.
  Arms: ACCESS

SUMMARY:
Aim is to test the effect of ACCESS ("Adaptive Computerized COPD Exacerbation Self-management Support"), a software application designed to support patients with COPD in self-management of exacerbations.

DETAILED DESCRIPTION:
Rationale: COPD exacerbations considerably affect patients' health status and contribute to COPD related costs. Patients often have problems in recognizing and responding promptly to exacerbations. Tools that support patients in exacerbation self-management such as paper exacerbation action plans and telemonitoring systems have shown some positive results on exacerbation related outcomes. However, many patients appear not to adhere to their action plan instructions. Besides, existing telemonitoring tools rely heavily on the input of healthcare professionals which makes it difficult to assess the true effects and cost effectiveness of telemonitoring systems.

Recently, the Radboud University has developed the "Adaptive Computerized COPD Exacerbation Self-management Support" (ACCESS) system. This software application integrates objective parameters, such as spirometry, pulse-oximetry, temperature, and self-reported symptom worsening into a Bayesian network model resulting in a weighted exacerbation risk prediction. Patients are able to monitor themselves at any given moment. The ACCESS system not only predicts whether an exacerbation is imminent, but also provides ad hoc tailored advice without interference of a healthcare professional.

Objective: In this project the primary aim is to assess the (cost-)effectiveness of the ACCESS system in the support of exacerbation self-management in patients with COPD.

Study design: A multicenter, pragmatic, two-arm, randomized controlled trial with a follow-up of 12 months per participant.

Study population: Patients with COPD, > 40 years old, with 2 or more self-reported symptom based exacerbations in the previous year.

Intervention: After a short self-management educational session on exacerbations, participants are randomized to either 1) exacerbation self-management support through the use of a paper exacerbation action plan (control group); or 2) exacerbation self-management support through the use of the ACCESS system (intervention group).

Participants in the intervention group are instructed to use ACCESS when they notice a change in COPD symptoms. Participants in the control group are instructed to use their paper action plan when they notice a change in COPD symptoms.

Main study parameters/endpoints:

Primary aim: to increase the number of exacerbation-free weeks. Secondary aims: to improve exacerbation self-management, exacerbation-management related self-efficacy, and quality of life. To decrease ER visits, hospital admissions and COPD related costs.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of COPD by spirometry (post-bronchodilator FEV1/FVC < 0.70);
* at least 2 self-reported exacerbations in the previous 12 months, i.e. a change for ≥ 2 consecutive days in either ≥ 2 major symptoms (dyspnea, sputum purulence, sputum amount) or any 1 major symptom plus any ≥ 1 minor symptoms (colds, wheeze, sore throat, cough).

Exclusion Criteria:

* severe co-morbid conditions that prohibit participation;
* unable to communicate in the Dutch language;
* difficulties using a smartphone;

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbation-free weeks | 1 year
  Measured with the Telephonic EXacerbation Assessment System (TEXAS) [Bischoff, ERJ, 2012]

SECONDARY OUTCOMES:
Improvement in exacerbation-related self-management behaviour | 1 year
  Prompt reaction and adequate response to symptoms, measured with the Telephonic EXacerbation Assessment System (TEXAS) [Bischoff, ERJ, 2012]
Improvement in Quality of Life | 1 year
  Measured with the Nijmegen Clinical Screening Instrument (NCSI)
Improvement in Quality of Life | 1 year
  Measured with the Clinical COPD Questionnaire (CCQ)
Improvement in Quality of Life | 1 year
  Measured with the Euroqol -5 dimensions (EQ-5d)
Improvement in self-efficacy | 1 year
  Measured with an exacerbation-related self-efficacy scale
Number of ER visits and hospital admissions | 1 year
  Measured with hospital and general practice medical records
Cost-effectiveness of ACCESS; ratio calculated with the use of medical records and questionnaires. | 1 year
  Costs consist of health care utilisation and patients' productivity losses, effectiveness is measured with EQ-5d.

CONTACTS AND LOCATIONS:
Overall Officials: Tjard Schermer, PhD, Principal Investigator — head of research unit
Locations (1):
- Radboud University Medical Centre, Department of Primary and Community Care, Nijmegen, Netherlands

REFERENCES:
- [Background] van der Heijden M, Lucas PJ, Lijnse B, Heijdra YF, Schermer TR. An autonomous mobile system for the management of COPD. J Biomed Inform. 2013 Jun;46(3):458-69. doi: 10.1016/j.jbi.2013.03.003. Epub 2013 Mar 15. PMID 23500485
- [Background] Bischoff EW, Boer LM, Molema J, Akkermans R, van Weel C, Vercoulen JH, Schermer TR. Validity of an automated telephonic system to assess COPD exacerbation rates. Eur Respir J. 2012 May;39(5):1090-6. doi: 10.1183/09031936.00057811. Epub 2011 Sep 15. PMID 21920893
- [Background] Bischoff EW, Hamd DH, Sedeno M, Benedetti A, Schermer TR, Bernard S, Maltais F, Bourbeau J. Effects of written action plan adherence on COPD exacerbation recovery. Thorax. 2011 Jan;66(1):26-31. doi: 10.1136/thx.2009.127621. Epub 2010 Oct 30. PMID 21037270
- [Background] van der Heijden M, Velikova M, Lucas PJ. Learning Bayesian networks for clinical time series analysis. J Biomed Inform. 2014 Apr;48:94-105. doi: 10.1016/j.jbi.2013.12.007. Epub 2013 Dec 18. PMID 24361389
- [Background] van der Heijden M, Lucas PJ. Describing disease processes using a probabilistic logic of qualitative time. Artif Intell Med. 2013 Nov;59(3):143-55. doi: 10.1016/j.artmed.2013.09.003. Epub 2013 Oct 7. PMID 24183893
- [Derived] Boer L, Bischoff E, van der Heijden M, Lucas P, Akkermans R, Vercoulen J, Heijdra Y, Assendelft W, Schermer T. A Smart Mobile Health Tool Versus a Paper Action Plan to Support Self-Management of Chronic Obstructive Pulmonary Disease Exacerbations: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Oct 9;7(10):e14408. doi: 10.2196/14408. PMID 31599729
- [Derived] Liu M, Stella F, Hommersom A, Lucas PJF, Boer L, Bischoff E. A comparison between discrete and continuous time Bayesian networks in learning from clinical time series data with irregularity. Artif Intell Med. 2019 Apr;95:104-117. doi: 10.1016/j.artmed.2018.10.002. Epub 2019 Jan 22. PMID 30683464